CLINICAL TRIAL: NCT00303056
Title: Efficacy and Safety of Intra-articular Multiple Doses of 500 µg Icatibant Including 40 mg Triamcinolone as Calibrator in a Randomized, Double-blind, Parallel-group, Placebo-controlled 13-week Multi-centre Study in Patients With Symptomatic Knee Osteoarthritis
Brief Title: Efficacy and Safety Study of Intra-articular Multiple Doses of Icatibant in Patients With Painful Knee Osteoarthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DRI6091; HOE140
Record Dates: First submitted 2006-03-14; First posted 2006-03-15 (Estimated); Last update posted 2012-02-17 (Estimated); Status verified 2012-02

CONDITIONS: Joint Disease
Keywords: Osteoarthritis; knee
MeSH Terms: conditions — Joint Diseases; Osteoarthritis | interventions — icatibant

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: HOE140 Icatibant

SUMMARY:
The primary objective is to compare the overall treatment effect on pain relief between icatibant and placebo. The secondary objectives are to assess the efficacy of icatibant in term of onset, extent and duration of pain relief relative to triamcinolone, to evaluate the safety of icatibant, to evaluate overall conditions of daily life after treatment with icatibant, to assess systemic exposure of icatibant following intra-articular injection.

DETAILED DESCRIPTION:
This is a multinational, randomized, placebo-controlled study to be conducted in Europe and the US. Study medication will be administered by intra-articular injection 3 times in weekly intervals, being followed by an observation period of further 11 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects with painful osteoarthritis of the knee.

Exclusion Criteria:

* Subjects presenting with diagnosis of OA < 3 months and an OA grading < K&L grade II, with any condition with impact on on the target indication, any test-compound-related condition, any study-related condition (all those conditions detailled in the CSP).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 590 (Actual)
Dates: Start 2006-02; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Pain during activity, at rest and at night will be measured daily via an electronic patient diary (EPD) using a 100-unit visual analog scale (VAS).

SECONDARY OUTCOMES:
Patient global assessment assessed daily as well as WOMAC scores at each visit and intake of rescue medication daily via EPD recording. Safety assessed at each visit and pharmacokinetics at visits 2, 3 & 4.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (5):
- Administrative Office, Bridgewater, New Jersey, United States
- Administrative Office, Vienna, Austria
- Administrative Office, Prague, Czechia
- Administrative Office, Berlin, Germany
- Administrative Office, Warsaw, Poland